CLINICAL TRIAL: NCT06422455
Title: Increasing Access to Genetic Testing in Underserved Patients Using a Multilingual Conversational Agent
Brief Title: Access to Genetic Testing in Underserved Patients With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Northeastern University (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19PS-24-3; NCI-2024-02187 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19PS-24-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH); R01CA263532 (NIH)
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Breast Carcinoma; Male Breast Carcinoma; Malignant Solid Neoplasm; Metastatic Prostate Carcinoma; Ovarian Carcinoma; Pancreatic Exocrine Neoplasm; Stage IVB Prostate Cancer American Joint Committee on Cancer v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Prostatic Neoplasms; Ovarian Neoplasms; Triple Negative Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Genetic Counseling; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Phase Arm A (PERLA) (Experimental): Patients receive access to PERLA comprising pre-test genetics education and standard post-test provider-based genetic counseling over 20-60 minutes. .
  Interventions: Other: Educational Intervention; Other: Electronic Health Record Review; Other: Genetic Counseling; Other: Interview; Other: Survey Administration
- Intervention Phase Arm B (usual care) (Active Comparator): Patients receive access to usual care pre- and post-test provider-based genetic counseling.
  Interventions: Other: Best Practice; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive provider-based genetic counseling
  Other Names: standard of care; standard therapy
  Arms: Intervention Phase Arm B (usual care)
Other: Educational Intervention — Receive genetics education
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Intervention Phase Arm A (PERLA)
Other: Electronic Health Record Review — Ancillary studies
Other: Genetic Counseling — Receive provider-based genetic counseling
  Arms: Intervention Phase Arm A (PERLA)
Other: Interview — Ancillary studies
  Arms: Intervention Phase Arm A (PERLA)
Other: Survey Administration — Ancillary studies

SUMMARY:
This study compares the experiences of people who receive information about genetic testing from a computer-generated character to patients who receive information from a human genetics healthcare provider. Patients with cancer are increasingly recommended for genetic testing as standard of care. Multiple factors contribute to low usage of genetic testing but for many patients the lack of access to genetic counseling and testing is an important and flexible factor. Lack of access is especially relevant to racial/ethnic minority patients and those living in non-metropolitan rural settings who are frequently cared for at safety-net hospitals with limited genetics services. Alternative delivery models are necessary to improve rates of access to genetic testing in patients with cancer. Health information technology is under used by genetics providers. A patient-facing relational agent (PERLA) will provide pre-test genetics education in both English and Spanish across two clinical settings to facilitate more timely access to genetic testing. Using the PERLA intervention may help researchers learn different ways to provide education about genetic testing to patients with cancer compared to usual care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain patient and provider input on the optimal content and format of a new relational agent (RA) intervention ("PERLA") for automated pre-test genetics education.

II. To obtain patient feedback on the usability of the English- and Spanish-language PERLAs.

III. To determine the acceptability of the newly designed English- and Spanish-language PERLAs among patients with cancer.

IV. To evaluate the impact of the English- and Spanish-language PERLAs on the proportion of patients who meet cancer-based genetic testing guidelines who receive genetic test results within 3 months of initiating cancer care.

V. To evaluate the potential barriers and facilitators to implementation of PERLA in the clinical setting.

OUTLINE:

DEVELOPMENT PHASE: Participants attend focus groups and provide feedback on the content, format, and usability of the PERLAs to enable to tailor the design of the intervention.

USABILITY PHASE: Participants attend usability testing and provide feedback through cognitive interviews.

PILOT TESTING PHASE: Participants evaluate the newly developed PERLAs and provide feedback through focused interviews and structured assessment.

INTERVENTION PHASE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive access to PERLA comprising pre-test genetics education and standard post-test provider-based genetic counseling over 20-60 minutes.

ARM B: Patients receive access to usual care pre- and post-test provider-based genetic counseling.

IMPLEMENTATION PHASE: Participants complete qualitative interviews to evaluate potential barriers and facilitators to implementation of PERLA in the clinic.

After completion of study intervention, patients are followed up at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diagnosed with least one of the following:

  * Epithelial ovarian cancer
  * Exocrine pancreatic cancer
  * Metastatic or high or very high-risk prostate cancer
  * Breast cancer at or before age 50
  * Bilateral breast cancer
  * Triple negative breast cancer
  * Male breast cancer OR
  * Healthcare provider who treats patients with any of the above types of cancer
* Able to read and write in English or Spanish
* Able to provide informed consent

Exclusion Criteria:

* Patients who cannot provide informed consent
* Patients who cannot see, read, or write
* Patients who have the cancer and clinical characteristics defined in the inclusion criteria, but who do not speak English or Spanish
* Patients with none of the listed cancer diagnoses and clinical characteristics
* Healthcare provider who do not treats cancer patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2027-10-24 (Estimated); Study Completion 2028-10-24 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who receive genetic testing | Up to 3 months
  The proportion of participants who receive genetic testing will be reported.

SECONDARY OUTCOMES:
Patient-reported outcomes | Up to 3 months
  Correlations with patient level factors, such as education, literacy, acculturation, and language will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Charite Ricker, MS, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Rochester, Rochester, New York